CLINICAL TRIAL: NCT03439527
Title: Open-label, Monocentric, First-in-man Trial to Assess Safety and Tolerability of a New Therapeutic Strategy for Stress Urinary Incontinence Based on the Implantation of Muscle Precursor Cells (MPCs)
Brief Title: Multisystem Cell Therapy for Improvement of Urinary Continence
Acronym: MUSIC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Hospital Tuebingen (Other); Salzburger Landeskliniken (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H2020-SC1-2016-2017; 731377 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2017-12-18; First posted 2018-02-20 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Urinary Stress Incontinence
Keywords: Muscle Precursor Cells
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — cyclic adenosine-5'-trimetaphosphate

STUDY DESIGN:
Intervention Model Description: Open-label, monocentric, first-in-man trial to assess safety and tolerability of a new therapeutic strategy for stress urinary incontinence based on the implantation of muscle precursor cells (MPCs) 40 female patients suffering from urinary incontinence since at least 6 months (predominant clinical diagnosis of SUI) and who are candidate for a surgical treatment will be included .
  All patients are treated by the same product: Autologous MPCs. After treatment, the patients will be randomized 1:1 in the MPC-group or NMES+MPC-group to investigate the benefits of an additional physiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPC-group (Experimental): All patients are treated by the same product: Autologous MPCs
  Interventions: Other: Muscle Precursor Cells (MPCs), ATMP
- NMES+MPC-group (Other): After treatment, the patients will be randomized 1:1 in the MPC-group or NMES+MPC-group to investigate the benefits of an additional physiotherapy (Neuromuscular Electromagnetic Stimulation, NMES)
  Interventions: Other: Muscle Precursor Cells (MPCs), ATMP

INTERVENTIONS:
Other: Muscle Precursor Cells (MPCs), ATMP — The advanced therapeutic investigational product, the MPCs, is a living, autologous cell-product isolated from a biopsy of the patient's own musculus soleus.

SUMMARY:
The rising success of cell therapies places an increasing burden on health care costs. Consequently, the need to reduce production costs while maintaining quality has been widely acknowledged. In addition, the demand for high-quality products with an optimal safety profile is increasing. The proposed cell treatment is the first therapeutical option with the possibility to revert the underlying condition. The investigators expect that this healing response will be achieved with minimal side effects justifying the addional costs and complexity.

DETAILED DESCRIPTION:
muscle precursor cells (MPCs) will be isolated from biopsies of the lower leg of patients, seeded, expanded and cultivated in vitro in a GMP facility to generate vital muscle cells dedicated for implantation.

These muscle cells exhibit myogenic phenotype (IHC and flow cytometry) and therefore morphological and histological prerequisites approximating the properties of native skeletal muscle tissue. The muscle progenitor cells shall be applied in external sphincter muscle for the treatment of patients with stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

Adult women 20y-60y

* Incontinence >/= grade I since at least 6 months
* Predominant clinical diagnosis of SUI
* Candidate for a surgical treatment (artificial urinary sphincter, synthetic compressive tapes or adjustable balloons).
* Post void residual volume of <100 ml (exclusion of overflow incontinence)
* Can independently use toilet without difficulty
* Capacity to answer the questionnaires of evaluation
* Negative blood test for: Human immunodeficiency virus (HIV 1/2), Hepatitis B HBsAg, Anti HBc, Hepatitis C Anti-HCV-Ab, Syphilis
* Competent to comprehend, sign and date informed consent form before any study-specific procedure is performed

Exclusion Criteria:

* History of anti-incontinence or prolapse surgery.
* Previous diagnosis of any of the following conditions, disorders, or diseases of the urinary tract:

  * Clinically significant cystocele or rectocele
  * Ureteric bladder, urethral or rectal fistula
  * Uncorrected congenital abnormality leading to urinary incontinence
  * Interstitial cystitis
* Urinary urgency that results in leakage (as a predominant symptom)
* Adult enuresis
* Urodynamically proven detrusor instability
* Sensory urgency defined as first sensation of bladder fill (urge to void) of <100 ml; bladder capacity of <300 ml
* No sensation at any time during the simple filling cystometry procedure
* Known urethral stenosis (ureterocystoscopy) or urethral diverticulum
* History of urogenital cancer or history of pelvic radiotherapy
* Women who are pregnant, breast feeding or <12 months postpartum Note: Female subjects who are surgically sterilized, hysterectomized or post-menopausal for longer than 2 years are not considered as having child bearing potential. No pregnancy test will be performed for this population.
* Untreated symptomatic urinary tract infection
* Fever (as defined by ≥ 38,5°C, axillar measurement), any infectious disease, cold or flu within the last 7 days
* Unstable severe systemic disease including uncontrolled hypertension, unstable angina, or myocardial infarction, severe coagulation disorders, bleeding diathesis, emboli, thrombophlebitis, infectious diseases, poor wound healing, and poorly controlled diabetes mellitus within 6 months before enrolment
* Any organic or psychiatric disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results.
* Known allergy or intolerance of at least one of the active ingredients or excipients of the investigational products
* Known allergy or intolerance of Penicillin or Streptomycin
* Known genetically determined or acquired muscular disease.
* Known Neurological disorder (Parkinson's disease, multiple sclerosis, spina bifida, medullary traumatism).
* Medication regimen including estrogens, anti-estrogens or diuretics where dose and/or frequency has not been stable for at least the past 12 weeks or is anticipated to change during the course of the study.
* Chronic use of any of the following drugs and not stopped for at least 2 weeks prior to inclusion into the study: selective serotonin and norepinephrine reuptake inhibitor antidepressant (SSNRI), alpha-receptor antagonists/agonists, beta-3-receptor agonists or anticholinergic/-muscarinic drugs.
* Chronic use of any of the following drugs and not stopped for at least 6 months prior to inclusion into the study: Antidepressants or neuroleptic drugs.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — due to injection technique
Enrollment: 10 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically relevant Adverse Events of MPCs or related to cell injection | at 3 months post-implantation
  Number of clinically relevant findings related to cell injection

SECONDARY OUTCOMES:
Feasibility of MPC injection | day of implantation
  Percentage of subjects with successful injection
Efficacy of MPC injection measured by post-void residual volume | at baseline, day of implantation, 1 month, 3 months and 6 months post-implantation
  post-void residual volume
Efficacy of MPC injection measured by Uroflowmetry | at baseline, day of implantation, 1 month, 3 months and 6 months post-implantation
  Uroflowmetry: urinary flow pattern
Efficacy of MPC injection measured by Urodynamic Evaluation | at baseline, 3 months and 6 months post-implantation
  2 Filling-Cystometries
Efficacy of MPC injection measured by Urodynamic Evaluation | at baseline, 3 months and 6 months post-implantation
  2 Pressure-Flow studies
Efficacy of MPC injection measured by Urodynamic Evaluation | at baseline, 3 months and 6 months post-implantation
  Urethal-Pressure-Profile
Efficacy of MPC injection measured by 1h pad test | at baseline, 1 month, 3 months and 6 months post-implantation
  1h pad test
Efficacy measured by average Incontinence Score | at baseline, 1 month, 3 months and 6 months post-implantation
  Incontinence Score. Range from 0 (no incentinence) to 21 (highly incontinent)
Efficacy measured by average score of Visual Analog Scale of degree of suffering | at baseline, 1 month, 3 months and 6 months post-implantation
  Visual Analog Scale of degree of suffering. Range 0 (worst) to 10 (best)
Efficacy measured by average score of Quality of Life | at baseline, 1 month, 3 months and 6 months post-implantation
  Quality of Life Score, using SF-36v2™ Health Survey
Efficacy | 6 months post-implantation
  Number for (planned) subsequent incontinence surgery
Number of patients with abnormal laboratory values and/or Adverse Events that are related to MPC injection | at baseline, day of implantation, 1 month, 3 months and 6 months post-implantation
  Safety measures (ultrasound, physical examination, laboratroy)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eberli, Prof, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No